CLINICAL TRIAL: NCT01119976
Title: Evaluation of the Association Between the Menstrual Cycle and Weight Loss in Healthy, Overweight Premenopausal Women
Brief Title: Association Between the Menstrual Cycle and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sierra Neuropharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0983
Record Dates: First submitted 2010-01-07; First posted 2010-05-10 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Reduced calorie diet and exercise plan that changes with phases of the menstrual cycle
  Interventions: Behavioral: Reduced calorie diet and exercise plan
- Group B (Active Comparator): Different reduced calorie diet and exercise plan based on MyPyramid.gov website
  Interventions: Behavioral: Different reduced calorie diet and exercise plan

INTERVENTIONS:
Behavioral: Reduced calorie diet and exercise plan — Participants will receive written diet and exercise instructions to follow for the duration of the study.
  Arms: Group A
Behavioral: Different reduced calorie diet and exercise plan — Participants will receive written diet and exercise instructions to follow for the duration of the study.
  Arms: Group B

SUMMARY:
This is a research study to look at the association between weight loss and the menstrual cycle in healthy, overweight, premenopausal women. Participants will be asked to follow a reduced-calorie diet and exercise plan for 3 months.

DETAILED DESCRIPTION:
Two different reduced calorie diet and exercise plans will be compared. One plan changes diet and exercise prescription with the phases of the menstrual cycle, while the other is a standard reduced calorie diet and exercise plan based on MyPyramid.gov website.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females between the ages of 18-40 (inclusive)
* BMI between 26.5-35.4 kg/m² (inclusive)
* Regular menstrual cycle (28 ± 3 days)
* Weight stable (within ± 3-kg) 2 months prior to study inclusion
* Must use barrier contraception (e.g. male/female condom) for the study's duration
* Must be willing to follow the prescribed diet/exercise plan for the study's duration

Exclusion Criteria:

* On hormonal contraceptives or any other daily use of medications which can make the subject unsuitable for inclusion in the study.
* Any significant health problem (history of cancer, HIV/AIDS, Diabetes, cardiovascular disease, untreated hypothyroidism, etc.)
* Restrictions against participating in cardiovascular exercise and strength training
* Any condition, which in the opinion of the investigator makes the subject unsuitable for inclusion in the study.
* Women who are pregnant, lactating, or planning to become pregnant during the study period

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months

SECONDARY OUTCOMES:
Waist Circumference | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James O Hill, Ph.D., Principal Investigator — University of Colorado Denver and Health Sciences Center
Locations (1):
- Center for Human Nutrition, Denver, Colorado, United States